CLINICAL TRIAL: NCT05433909
Title: Microbiota and Immunoassay in Women With and Without Endometriosis: a Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Direzione Ginecologia, Principal Investigator, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 0009206 u
Record Dates: First submitted 2022-03-09; First posted 2022-06-27 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Endometriosis; Endometriosis-related Pain
Keywords: Diagnosis; Microbiota; immunoassay
MeSH Terms: conditions — Endometriosis; Disease | interventions — Blood Specimen Collection; Defecation

STUDY DESIGN:
Intervention Model Description: Biological non-pharmacological Pilot study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endometriosis group (Experimental): The endometriosis group will include women who will undergo surgery for endometriosis.
  Interventions: Diagnostic Test: Blood, fecal, vaginal and endometrial liquid samples
- Control Group (Experimental): The control group include women who will undergo surgery for other gynecological diseases in which the presence of endometriosis will be excluded during the operation.
  Interventions: Diagnostic Test: Blood, fecal, vaginal and endometrial liquid samples

INTERVENTIONS:
Diagnostic Test: Blood, fecal, vaginal and endometrial liquid samples — During the surgical pre-hospitalization, eligible patients who accept participation in the study will undergo a blood sample and collection of stool samples.
  Before surgery, after anesthesia, they will undergo a vaginal swab and endometrial fluid sampling.

SUMMARY:
Endometriosis is an estrogen-dependent chronic inflammatory disease characterized by the presence of endometrial tissue outside the uterine cavity. This pathology has a prevalence of about 5-10% in reproductive-aged women. Endometriosis therapy uses two options: surgical or medical (hormonal) but none can be considered completely resolving. Related signs and symptoms include dysmenorrhea, dyspareunia, infertility, dysuria and dyschezia. In addition to typical gynecological symptoms, gastrointestinal symptoms (bloating, nausea, constipation, diarrhea and vomiting) affect up to 90% of patients with endometriosis. Despite its high prevalence and associated morbidity, its etiology is still unclear and is thought to be multifactorial, and genetic, hormonal, environmental and immunological factors contribute to it. Several studies have shown a significant association between abnormal immune response and maintenance of disease activity in women with endometriosis.

The microbiome contains all the genetic material of microbes, including bacteria, fungi, viruses and Archaea, which live inside the host and regulate various physiological functions. The set of these bacteria, fungi, viruses and Archaea is called a microbiota. The influence of the microbiome on immunomodulation and the development of various inflammatory diseases is well established. Conversely, little is known about the presence and composition of the microbiome in the female reproductive system and its role in the development of endometriosis or other gynecological conditions. Considering the altered inflammatory state typical of endometriosis, it seems logical to postulate a potential role of the microbiome in the etiopathogenesis of this pathology. Interestingly, the microbiome affects estrogen metabolism and estrogen affects the gut microbiome. Since endometriosis is an estrogen-dependent disease, a picture of intestinal dysbiosis resulting in abnormal circulating estrogen levels could potentially contribute to the development of this disease.

ELIGIBILITY:
Inclusion Criteria:

* BMI <30 kg / m2
* no hormonal therapy (estrogen-progestin, progestogen, GnRH analogues) in progress for at least 1 month
* the endometriosis group include women who will undergo surgery for endometriosis. The control group include women who will undergo surgery for other gynecological indications (i.e .: abdominal surgical emergencies, tubal infertility, non-endometriotic ovarian cysts) in which the presence of endometriosis will be excluded during the surgery.

Exclusion Criteria:

* hormonal therapy in progress (estrogen-progestins, progestins, GnRH analogues)
* antibiotic and / or probiotic therapy in the 8 weeks before the samples
* pregnancy
* menopausal state
* BMI ≥ 30 kg / m2
* presence of active systemic diseases, neoplasms, positive clinical history for autoimmune diseases, active vaginosis or positive history for pelvic inflammatory disease

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-04-09 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Intestinal, vaginal and endometrial microbiota in patients with and without endometriosis | 8 months
  The intestinal, vaginal and endometrial microbiota in patients with endometriosis is different than the intestinal, vaginal and endometrial microbiota in patients without endometriosis
inflammatory, immunophenotype and hormonal status in patients with and without endometriosis | 8 months
  Differences of the inflammatory state, immunophenotype and hormonal status of the two groups of patients.

SECONDARY OUTCOMES:
Molecular, immunological characteristics of the inflammatory endometriosis environment | 8 months
  the molecular and immunological characteristics of the inflammatory environment of endometriotic lesions and peripheral blood changed from women with and without endometriosis
Microbiota and sites, symptoms, hormonal treatments of endometriosis | 8 months
  Any differences regarding the composition of the microbiota based on the location of the disease, the presence of symptoms or previous hormonal treatments.
The impact of the various factors in determining the disease | 8 months
  The relative impact of the various factors in determining the disease combining characteristics of the microbiota with clinical data (genetic, serological, immunological and metabolic).

CONTACTS AND LOCATIONS:
Overall Officials: Laura Buggio, MD, Principal Investigator — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Locations (1):
- Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico, Milan, Italy

IPD SHARING:
Plan to Share IPD: No